CLINICAL TRIAL: NCT00845897
Title: Botulinum Toxin Effects on Plantar Ulcer Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mary Hastings, PT, DPT, ATC, Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 04-0493; R21HD048972 (NIH)
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Results first posted 2012-02-02 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus; Peripheral Neuropathy; Plantar Ulcers
Keywords: Diabetes mellitus; plantar ulcers; peripheral neuropathy
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases; Foot Ulcer | interventions — Botulinum Toxins; Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo (saline) injections into 6 sites in the calf muscle
  Interventions: Drug: Saline
- 2 (Active Comparator): Total 200 units of Botulinum Toxin injected into 6 sites into the calf muscles.
  Interventions: Drug: Botulinum Toxin
- 3 (Active Comparator): 300 units of botulinum toxin injected into 6 sites in the calf muscle
  Interventions: Drug: Botulinum Toxin

INTERVENTIONS:
Drug: Botulinum Toxin — 200 units of botulinum toxin, and 300 units of botulinum toxin. Injection are given at one session. 2 injections into the medial gastrocnemius, 2 injections into the lateral gastrocnemius, and 2 injections into the soleus
  Other Names: botox
  Arms: 2; 3
Drug: Saline — Placebo (saline) (3cc). Injection are given at one session. 2 injections into the medial gastrocnemius, 2 injections into the lateral gastrocnemius, and 2 injections into the soleus
  Arms: 1

SUMMARY:
The purpose of this grant is to collect pilot data to assess the amount of botulinum toxin that needs to be injected into the calf muscles of subjects with diabetes mellitus, peripheral neuropathy, and a plantar ulcer to decrease muscle strength. We hypothesize that a decrease in plantar flexor muscle strength will temporarily decrease plantar pressure. The decrease in plantar pressure will provide temporary protection to the new tissue as it gains tolerance to high stress with the long term potential outcome as a decrease in the ulcer recurrence rate.

DETAILED DESCRIPTION:
Please read "Brief Summary"

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of diabetes mellitus and determination of diminished or absent plantar sensation
* A recurrent forefoot plantar ulcer; at least the second occurrence of a plantar ulcer or a previous failure to heal a plantar ulcer with reasonable treatment intervention (Total contact casting, off loading boot, molded ankle foot orthotic, Gillette, or therapeutic footwear modifications)
* Ambulatory

Exclusion Criteria:

* Active infection in the involved foot
* Previous botulinum toxin injections
* Ulcers on the dorsal surface of the foot
* Ankle-brachial index <0.45
* History of cerebral vascular accident or other neurological problems complicating their rehabilitation
* Women of childbearing years unless pregnancy test is agreed upon, completed, and negative and agree to use some form of contraception during the study.
* Current drug therapy that includes an anticoagulant
* History of a neuromuscular disease, except peripheral neuropathy as a result of diabetes mellitus

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary K Hastings, PT, DPT, ATC, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Placebo (saline) injections into 6 sites in the calf muscle
- 200 Units of Botox: Total 200 units of Botulinum Toxin injected into 6 sites into the calf muscles.
- 300 Units of Botox: 300 units of botulinum toxin injected into 6 sites in the calf muscle
Period: Overall Study
Arm/Group | Placebo Group | 200 Units of Botox | 300 Units of Botox
Started | 5 | 7 | 5
Completed | 3 | 2 | 2
Not Completed | 2 | 5 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 3 | 2
Not completed — Ulcer did not heal | 1 | 0 | 1
Not completed — Too ill to participate | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | 200 Units of Botox | 300 Units of Botox | Total
Number analyzed (Participants) | 5 | 7 | 5 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 4 | 15
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 14
  Male | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Plantar Flexor Muscle Strength
Description: Concentric plantar flexor torque was assessed using the Biodex System 3 Pro Orthopedic Testing & Rehabilitation dynamometer. Plantar flexor peak torque was measured at 60 deg/sec, which is comparable to the angular velocity of the ankle joint during the stance phase of walking. Three trials of each foot were completed. Peak torque was calculated as the average of the two highest torque values across trials and results were expressed as Nm. A positive value represents an increase in torque while a negative value represents a decrease in torque.
Time Frame: Pre-treatment, 2 weeks after injection, upon ulcer healing, 3 months and 6 months after ulcer healing
Measure: Mean (Standard Deviation); unit: Plantar Flexor Torque (Nm)
Groups:
- Botulinum Toxin 200 Units: 200 units of Botox®
- Placebo: Saline
- Botulinum Toxin 300 Units: 300 units of Botox®
Arm/Group | Botulinum Toxin 200 Units | Placebo | Botulinum Toxin 300 Units
Number analyzed (Participants) | 7 | 5 | 5
Plantar Flexor Torque (Nm) | -8 (11) | 3 (4) | 6 (10)

2. Secondary Outcome: Barefoot Plantar Pressure
Description: Novel emed pressure platform was used for data collection. A two-step method of data collection was used and a minimum of two trials of each foot were recorded. The plantar pressure map was divided into 3 horizontal masks using Percent Mask software and peak plantar pressure was determined for the forefoot region. Results are expressed in N/cm^2.
Time Frame: pre-injection, 2 weeks post injection, post healing, and 3 and 6 months post healing
Measure: Mean (Standard Deviation); unit: Peak Plantar Pressure (N/cm^2) changes
Arm/Group | Botulinum Toxin 200 Units | Placebo | Botulinum Toxin 300 Units
Number analyzed (Participants) | 7 | 5 | 5
Peak Plantar Pressure (N/cm^2) changes | -4 (16) | 0 (11) | 0 (5)

ADVERSE EVENTS:
Arm/Group | Placebo Group | 200 Units of Botox | 300 Units of Botox
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No